CLINICAL TRIAL: NCT04840446
Title: Evaluation of Modified Adhesives With Dexcom G6 Sensor
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: PTL-904288
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Diabetes
Keywords: Diabetes; Continuous Glucose Monitoring Systems
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Dexcom Continuous Glucose Monitoring System — Dexcom Sensor

SUMMARY:
The purpose of the study is to collect and compare information on the performance of CGM adhesives in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. No previously self-reported adhesive reactions to the any continuous glucose monitor (CGM);

Exclusion Criteria:

1. Extensive skin changes/diseases that preclude wearing the required number of devices (e.g., history of severe reactions from adhesive wear, extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
2. Current or anticipated use of systemic corticosteroids (oral, injectable, or intravenous)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be identified via diabetes patient website and/or virtual registry.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Adhesiveness and survivability of the adhesives | 10-days
  Number of adhesives that survive on the body during wear period

SECONDARY OUTCOMES:
Skin irritation with the adhesives | 10-days
  Proportion of participants who self-report skin irritation during wear period.
Occurrence of adverse events with the adhesives | 10-days
  Highest Draize scale score for adhesive erythema, and edema during wear period. Recorded medical adhesive-related skin injuries (MARSI) and severity during wear period.
Assess user preference or acceptance of the adhesives worn during the study | 10-days
  Final day post-study satisfaction questionnaire (for each adhesive) will be given a score by taking the mean response on the scale 1-5. Satisfaction scores will be tabulated by adhesive.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Mouse, BS, Principal Investigator — Jaeb Center for Health Research
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No